CLINICAL TRIAL: NCT00511758
Title: Pilot Study of a Digital Imaging Aid for Assessment of Cervical Dysplasia
Brief Title: Digital Imaging Aid for Assessment of Cervical Dysplasia
Status: Terminated | Type: Observational
Why Stopped: Low accrual rate.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2007-0230
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Cervical Dysplasia
Keywords: Cervical Dysplasia; Digital Imaging; Colposcopy; Cervix
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Quantitative Phase Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Digital Imaging Device: Patients with a diagnosis of cervical dysplasia that are scheduled for a colposcopy.
  Interventions: Procedure: Digital Imaging

INTERVENTIONS:
Procedure: Digital Imaging — Images of the cervix will be taken using different types of light and compared with the colposcopy procedure.

SUMMARY:
The overall objective of this study is to evaluate whether polarized or green filtered digital imaging can assist clinicians to screen for premalignant lesions in the cervix.

The specific aims of the study are:

* To compare polarized and green filtered digital images of the cervix, to standard white light images, colposcopic evaluation and to pathologic analysis of biopsied tissue.
* To develop algorithms to discriminate between normal and abnormal tissue based on digital images of the cervix.
* To analyze digital images to determine which types of optical information yield the most diagnostically useful data.

DETAILED DESCRIPTION:
If you agree to take part in this study, digital imaging will be performed for research purposes, after your routine colposcopy of your cervix.

VISUAL DETECTION OF PRECANCEROUS LESIONS:

Reflectance (the ability of an area to reflect light) imaging helps doctors visually tell the difference between precancerous tissue, cancerous tissue, and normal tissue in the cervix. Researchers want find out whether a digital camera image can be as effective as colposcopy at screening for precancerous tissue.

STUDY PARTICIPATION:

You will be seen in the clinic during a routine visit. Your cervix will first be examined by the clinician using a standard white light headlamp, and the image will be recorded.

Your cervix will then be re-examined with the digital camera, which will involve the use of different types of light (standard white light, green filtered light, cross and parallel polarized light). These digital images will be taken before and after acetic acid (vinegar) is applied.

Researchers will use these images to make comparison studies with the colposcopy procedure.

LENGTH OF STUDY:

Your participation will be finished on this study once your cervix has been examined with the digital camera.

This is an investigational study. Up to patients 20 will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older who are referred to the University of Texas MD Anderson Cancer Center Colposcopy Clinic for colposcopy are eligible for this study.
* Patients must sign an informed consent indicating awareness of the investigational nature of this study.

Exclusion Criteria:

* Patients who are pregnant are not eligible for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of cervical dysplasia that are scheduled for a colposcopy.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2007-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Evaluate whether a digital camera image can work as well as colposcopy at detecting precancerous tissue. | 2 Year

CONTACTS AND LOCATIONS:
Overall Officials: Michele Follen, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org